CLINICAL TRIAL: NCT06819579
Title: Exploring the Optimal Concentration of Lidocaine Test Dose for Labor Analgesia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Bing Chen, Ph.D, Professor Bing Chen, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024.276
Record Dates: First submitted 2025-01-24; First posted 2025-02-11 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-02

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1.5% Lidocaine (Active Comparator): After successful epidural puncture, 3ml of 1.5% lidocaine was injected as a test dose
  Interventions: Drug: 1.5% Lidocaine
- 1.0% Lidocaine (Experimental): After successful epidural puncture, 5ml of 1% lidocaine was injected as a test dose
  Interventions: Drug: 1.0% Lidocaine
- 0.5% Lidocaine (Experimental): After successful epidural puncture, 10ml of 0.5% lidocaine was injected as a test dose
  Interventions: Drug: 0.5% Lidocaine

INTERVENTIONS:
Drug: 1.5% Lidocaine — After successful epidural puncture, 3ml of 1.5% lidocaine was injected as a test dose
  Other Names: Lidocaine
  Arms: 1.5% Lidocaine
Drug: 1.0% Lidocaine — After successful epidural puncture, 5ml of 1% lidocaine was injected as a test dose
  Arms: 1.0% Lidocaine
Drug: 0.5% Lidocaine — After successful epidural puncture, 10ml of 0.5% lidocaine was injected as a test dose
  Arms: 0.5% Lidocaine

SUMMARY:
This study aims to compare the analgesia effects and side effects of different concentrations of test dose lidocaine (1.5% lidocaine 3 ml, 1.0% lidocaine 5 ml, 0.5% lidocaine 10 ml) in labor analgesia, so as to provide a scientific basis for the clinic al practice of labor analgesia.

DETAILED DESCRIPTION:
Epidural analgesia is the most effective and widely used analgesic method for relieving labor pain in clinical practice. However, inadvertent insertion of an epidural catheter into a blood vessel or subarachnoid space may result in local anesthesia or total spinal anesthesia, which can be life-threatening. Therefore, a low-concentration, low-volume dose of local anesthetic is usually injected as a test dose before injecting a large dose of local anesthetic through the epidural catheter to ensure that the catheter is within the epidural space. At present, the guidelines recommend 3 ml of 1.5% lidocaine as the test dose, but in clinical practice and the study of Chen et al., it was found that the test dose of 1.5% lidocaine 3ml still has a high incidence of lower limb motor block of 57.1%, which affects maternal activity and labor progression. In addition, Liu Henry et al. found that the incidence of 0.5% lidocaine 10 ml test dose-induced motor block was 0%, and the analgesic effect could be quickly achieved. Therefore, it is uncertain which concentration of lidocaine has the fastest onset of analgesia and the fewest side effects in labor analgesia. Therefore, this study aims to compare the effects of different concentrations of lidocaine (1.5% lidocaine 3 ml, 1.0% lidocaine 5 ml, 0.5% lidocaine 10 ml) in labor analgesia, so as to provide a scientific basis for the clinical practice of labor analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton primipara
2. Aged 20-40 years
3. Pre-assessed as eligible for vaginal delivery
4. Height between 155-170 cm, BMI between 18.5-35 kg/m²
5. Cervical dilation between 2-6 cm
6. No significant history of cardiopulmonary disease
7. No history of surgical trauma
8. American Society of Anesthesiologists (ASA) Grades I-III
9. Patients are willing to participate and be able to understand and sign an informed consent form

Exclusion Criteria:

1. Contraindications for spinal anesthesia, such as coagulopathy or ongoing anticoagulant therapy, infection at the puncture site, bacteremia, epidural abscess, increased intracranial pressure, severe hypovolemia
2. Physical or mental disabilities, such as scoliosis and depression, alcohol or drug abuse
3. Major organ diseases, such as hyperthyroidism, cardiopulmonary diseases, diabetes treated with insulin, and neuromuscular diseases
4. Numerical Pain Rating Scale (NPRS) < 5
5. Refusal to participate in the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of motor block | 3,5,7,9,11,13,15,20,25,30 minutes after lidocaine administration
  Bromage Scores were used to grade movement block: I free movement of legs and feet, II free movement of feet with only bent knees, III free movement of feet without bending knees, IV no movement of legs and feet, with scores of II, III and IV considered as movement block.

SECONDARY OUTCOMES:
Pain scores | 3,5,7,9,11,13,15,20,25,30 minutes after lidocaine administration
  Pain scores is assessed by the Numerical Pain Rating Scale (NPRS, where 0 means no pain and 10 means no pain tolerance)
Time of analgesia onset | 3,5,7,9,11,13,15,20,25,30 minutes after lidocaine administration
  Pain scores is assessed by the Numerical Pain Rating Scale (NPRS, where 0 means no pain and 10 means no pain tolerance). Analgesia is considered effective when NPRS is ≤3 or NPRS is reduced by ≥ 50% of the baseline value.
Sensory block level | 3,5,7,9,11,13,15,20,25,30 minutes after lidocaine administration
  Midabdominal line acupuncture was used to assess the sensory block level
Incidence of complications related to labor analgesia | 30 minutes after lidocaine administration
  Ask the patient if they have discomfort such as leg warmth, leg numbness, trembling, itching, headache, tinnitus, etc.
frequency and intensity of uterine contractions | 30 minutes after lidocaine administration
  A contraction monitor is used to monitor the intensity and frequency of contractions
Maternal blood pressure | 5,10,15,20,25,30 minutes after lidocaine administration
  Automated monitoring with an ECG monitor
Maternal heart rate | 5,10,15,20,25,30 minutes after lidocaine administration
  Automated monitoring with an ECG monitor
Pulse oximetry （SPO2） | 5,10,15,20,25,30 minutes after lidocaine administration
  Automated monitoring with an ECG monitor
fetal heart rate | 5,10,15,20,25,30 minutes after lidocaine administration
  Automatically monitored using a fetal heart rate monitor
Patient satisfaction score | 30 minutes after lidocaine administration
  Numerical rating scale was used to score (0, completely dissatisfied; 1. Neutral; 2, satisfaction; 3, completely satisfied)
First stage of labor | From enrollment to 1 minute after the baby comes out.
  The first stage of labor begins when labor starts and ends with full cervical dilation to 10 centimeters.
Second stage of labor | From enrollment to 1 minute after the baby comes out.
  The time from the cervix dilated to 10 centimeters to the baby comes out.
neonatal Apgar score | 1, 5, and 10 minutes after baby comes out.
  The Apgar score is to evaluate the presence or absence of neonatal asphyxia and the severity of asphyxia from five aspects: Appearance, Pulse, Grimace, Activity and Respiration after birth, with each item being 0~2 points and a full score of 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Chen, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available with the responding author when required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available when publish and keep it for 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal.